CLINICAL TRIAL: NCT02578368
Title: Effect of Chemotherapy Alone vs. Chemotherapy Followed by Surgical Resection on Survival and Quality of Life in Patients With Limited-metastatic Adenocarcinoma of the Stomach or Esophagogastric Junction - A Phase III Trial of Arbeitsgemeinschaft Internistische Onkologie/Chirurgische Arbeitsgemeinschaft Onkologie/Chirurgische Arbeitsgemeinschaft für Den Oberen Gastrointestinaltrakt (AIO/CAO-V/CAOGI)
Brief Title: Chemotherapy Alone vs. Chemotherapy + Surgical Resection in Patients With Limited-metastatic Adenocarcinoma of the Stomach or Esophagogastric Junction
Acronym: FLOT5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Krankenhaus Nordwest (Other)
Collaborators: German Research Foundation (Other); Arbeitsgemeinschaft fur Internistische Onkologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RENAISSANCE
Record Dates: First submitted 2015-10-12; First posted 2015-10-16 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; perioperative; FLOT; limited metastatic; GEJ cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Docetaxel; Trastuzumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: FLOT chemotherapy + surgery (OP) (Experimental): 4 cycles (8 weeks) FLOT pre-OP - surgery - 4-8 cycles FLOT (8-16 weeks) post-OP
  Docetaxel (50 mg/m2) in 250 ml sodium chloride (NaCl) 0.9% i.v. for 1 h, d1; Oxaliplatin (85 mg/m2) in 500 ml G5% (glucose 5%) i.v. for 2 h, d1; Leucovorin (Ca-folinate) (200 mg/m2) in 250 ml NaCl 0.9% i.v. for 1 h, d1*; 5-FU (2600 mg/m2) continuous infusion for 24 h, d1; Repeated every two weeks (qd15).
  * Leucovorin can be replaced by sodium folinate. Dose adjustment necessary if levo-leucovorin is used instead of racemic leucovorin mixture.
  For HER-2 positive disease, trastuzumab should be added:
  Trastuzumab 4 mg/kg body weight (6 mg loading dose at 1st administration), i.v. for 1 h, d1
  For PD-L1 positive disease (CPS ≥ 5), nivolumab can be added according to SmPC:
  Nivolumab 240 mg i.v. for 30 min, d1, repeated every two weeks (q15d)
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Docetaxel; Drug: Trastuzumab; Drug: sodium folinate; Procedure: Surgery
- Arm B: FLOT chemotherapy alone (Active Comparator): 4 cycles (8 weeks) FLOT followed by further 4-8 cycles FLOT (8-16 weeks)
  Docetaxel (50 mg/m2) in 250 ml sodium chloride (NaCl) 0.9% i.v. for 1 h, d1; Oxaliplatin (85 mg/m2) in 500 ml G5% (glucose 5%) i.v. for 2 h, d1; Leucovorin (Ca-folinate) (200 mg/m2) in 250 ml NaCl 0.9% i.v. for 1 h, d1*; 5-FU (2600 mg/m2) continuous infusion for 24 h, d1; Repeated every two weeks (qd15).
  * Leucovorin can be replaced by sodium folinate. Dose adjustment necessary if levo-leucovorin is used instead of racemic leucovorin mixture.
  For HER-2 positive disease, trastuzumab should be added:
  Trastuzumab 4 mg/kg body weight (6 mg loading dose at 1st administration), i.v. for 1 h, d1
  For PD-L1 positive disease (CPS ≥ 5), nivolumab can be added according to SmPC:
  Nivolumab 240 mg i.v. for 30 min, d1, repeated every two weeks (q15d)
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Docetaxel; Drug: Trastuzumab; Drug: sodium folinate

INTERVENTIONS:
Drug: 5-Fluorouracil — 2600 mg/m², d1 i.v., every 2 weeks
  Other Names: 5-FU
Drug: Leucovorin — 200 mg/m², d1, i.v., every 2 weeks
  Other Names: calcium folinate
Drug: Oxaliplatin — 85 mg/m², d1, i.v., every 2 weeks
Drug: Docetaxel — 50mg/m², d1, i.v., every 2 weeks
Drug: Trastuzumab — 4 mg/kg BW (6 mg loading dose at 1st administration), i.v. for 1 h, d1, i.v., every two weeks
Drug: sodium folinate — can be used to replace leucovorin (calcium folinate)
Procedure: Surgery — Aim of surgical resection is a complete (R0) resection of the primary tumor and the metastases or a complete macroscopic cytoreduction of the metastases.
  Arms: Arm A: FLOT chemotherapy + surgery (OP)

SUMMARY:
Previously untreated patients with limited metastatic stage (see protocol for details on criteria) will receive 4 cycles of FLOT (5-Fluorouracil, Leucovorin, Oxaliplatin and Docetaxel). Patients without disease progression will be randomized 1:1 to receive additional chemotherapy cycles (4-8 cycles of FLOT) or surgical resection followed by subsequent chemotherapy (4-8 cycles of FLOT). Main objective of the study is overall survival. Most important secondary objective is the quality of life under treatment and during follow-up.

DETAILED DESCRIPTION:
Patients with potentially limited metastatic gastric cancer or adenocarcinoma of the gastroesophageal junction (GEJ) potentially fulfilling the selection criteria and who gave informed consent will undergo a careful screening and a central review process. 271 patients are to be allocated to the trial, of which at least 176 patients will be randomized. The primary objective is to extend overall survival, while preserving quality of life. The study has an 80% power to detect a statistically significant improvement (hazard ratio, HR 0.65) in overall survival in favor of the bimodal strategy. Quality of life (QoL) under treatment and during follow-up represents the most important secondary endpoint.

All patients enrolled will receive four cycles (= 8 weeks) of FLOT. For HER-2 (human epidermal growth factor receptor 2) positive disease, trastuzumab should be added.

After the 4th cycle of FLOT, patients will undergo a repeated imaging (esophago-gastro-duodenoscopy, CT/MRI or PET scan of the involved organs). Patients with disease progression will be taken out of the trial. Patients with stable disease, partial or complete remission will be stratified by tumor location (gastric vs. GEJ adenocarcinoma), response to preoperative FLOT (complete or partial remission vs. stable disease) and based on whether they have distant lymph node metastases only or additional organ involvement and will be randomized 1:1 to Arm A (with surgery) or B (no surgery).

Arm A:

Surgery will be scheduled 4-6 weeks after d1 of the last cycle of preoperative chemotherapy (d1 + 4-6 weeks). The protocol gives detailed recommendations for resection of the primary tumor as well as the metastases. Post-operatively, further 4-8 cycles of FLOT can be administered.

Arm B:

Patients will be treated with additional 4-8 cycles of FLOT. Surgical interventions are allowed for palliation.

In both of the arms, tumor assessments (CT/MRI or PET of the relevant organs) are performed prior to randomization and then every 3 months thereafter until progression/relapse, death or end of follow-up.

Quality of life (QoL) will be assessed at baseline, prior to randomization, and every 3 months after randomization during treatment and in the follow-up phase, together with tumor assessments.

Survival status and status on relapse/first progress of disease will be assessed every 3 months for up to 5 years after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed limited metastatic gastric or GEJ adenocarcinoma.*
2. Medical and technical operability of the primary.
3. Metastatic lesions are resectable or can be controlled by local ablative procedure (central evaluation).
4. No prior chemotherapy and no prior tumor resection.
5. Female and male patients ≥ 18 years. Patients in reproductive age must be willing to use adequate contraception during the study and 3 months after the end of the study (appropriate contraception is defined as surgical sterilization (e.g., bilateral tubal ligation, vasectomy), hormonal contraception (implantable, patch, oral), and double-barrier methods (any double combination of: intrauterine device, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap)). Female patients with childbearing potential need to have a negative pregnancy test within 7 days before study start.
6. ECOG (Eastern Cooperative Oncology Group) Performance Status 0 or 1
7. Adequate hematological, hepatic and renal function parameters:

   * Leukocytes ≥ 3000/µl
   * Platelets ≥ 100,000/µl
   * Serum creatinine ≤ 1.5 x upper limit of normal, or glomerular filtration rate (GFR) > 40 ml/min
   * Bilirubin ≤ 1.5 x upper limit of normal
   * AST (aspartate aminotransferase) and ALT (alanine transaminase) ≤ 3.5 x upper limit of normal
   * Alkaline phosphatase ≤ 6 x upper limit of normal
8. Written informed consent of the patient.

(*) Definition of the limited metastatic status is:

1. Retroperitoneal lymph node metastases (RPLM) (e.g., para-aortal, intra-aorto-caval, parapancreatic or mesenterial lymph nodes) only (Note: in duodenum invading gastric cancer, retropancreatic nodes are not regarded M1) or/and
2. at maximum one organ involved with or without RPLM according to the following schema: I. Localized potentially operable peritoneal carcinomatosis: stage P1 according to classification of the "Japanese Research Society for Gastric Cancer" (Clinically visible carcinomatosis of the peritoneum or of the pleura and >P1 peritoneal carcinomatosis are not allowed!) or II. Liver: maximum of 5 metastatic lesions that are potentially resectable or III. Lung: unilateral involvement, potentially resectable or IV. Uni- or bilateral Krukenberg tumors (ovarian met.) in the absence of macroscopic peritoneal carcinomatosis or V. Uni- or bilateral adrenal gland metastases or VI. Extra-abdominal lymph node metastases such as supraclavicular or cervical lymph node involvement or VII. Localized bone involvement (defined as being within one radiation field) or VIII. Other metastatic disease location that is considered limited by the investigator and is confirmed by the review committee

Exclusion Criteria:

1. Medical inoperability
2. Inability to understand the aims of the study and/or protocol procedures
3. Metastatic disease not fulfilling the criteria of limited disease mentioned in the inclusion criteria or non-metastatic stage (cM0)
4. Cirrhosis of the liver, pronounced alcohol abuse with anticipated detoxification, severe pulmonary infection with considerable reduction of pulmonary function
5. Primary not resectable
6. Hypersensitivity to 5-fluorouracil, leucovorin, oxaliplatin, or docetaxel
7. Contraindication versus 5-fluorouracil, leucovorin, oxaliplatin, or docetaxel (see specific product information)
8. Clinically significant active coronary heart disease, cardiomyopathy or congestive heart failure, NYHA (New York Heart Association) III-IV
9. Clinically significant valvular defect
10. Past or current history of other malignancies unless curatively treated and without evidence of disease for more than 3 years, except for curatively treated basal cell carcinoma of the skin and in situ carcinoma of the cervix
11. Known brain metastases
12. Other severe internal disease or acute infection
13. Peripheral polyneuropathy > NCI grade II
14. Serious hepatic impairment (AST/ALT>3.5xULN, AP>6xULN, bilirubin>1.5xULN; ULN = upper limit of normal)
15. Chronic inflammatory bowel disease
16. Any other concurrent antineoplastic treatment including irradiation
17. Participation in another clinical study
18. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 5 years follow-up

SECONDARY OUTCOMES:
Quality of life (QoL) adjusted OS | up to 5 years follow-up
QoL-response | up to 5 years follow-up
QoL mean scores | up to 5 years follow-up
OS in patients with lymph node metastases only | up to 5 years follow-up
Progression free survival (PFS) | up to 5 years follow-up
Surgical morbidity | up to 2 months after surgery
Surgical mortality | up to 2 months after surgery
Toxicity - Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From signature of the informed consent form (ICF) up to 30 days after last administration

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, MD, Study Director — Institute of Clinical Cancer Research (IKF), Krankenhaus Nordwest; University Cancer Center Frankfurt (UCT)
Locations (1):
- Krankenhaus Nordwest, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Derived] Al-Batran SE, Goetze TO, Mueller DW, Vogel A, Winkler M, Lorenzen S, Novotny A, Pauligk C, Homann N, Jungbluth T, Reissfelder C, Caca K, Retter S, Horndasch E, Gumpp J, Bolling C, Fuchs KH, Blau W, Padberg W, Pohl M, Wunsch A, Michl P, Mannes F, Schwarzbach M, Schmalenberg H, Hohaus M, Scholz C, Benckert C, Knorrenschild JR, Kanngiesser V, Zander T, Alakus H, Hofheinz RD, Roedel C, Shah MA, Sasako M, Lorenz D, Izbicki J, Bechstein WO, Lang H, Moenig SP. The RENAISSANCE (AIO-FLOT5) trial: effect of chemotherapy alone vs. chemotherapy followed by surgical resection on survival and quality of life in patients with limited-metastatic adenocarcinoma of the stomach or esophagogastric junction - a phase III trial of the German AIO/CAO-V/CAOGI. BMC Cancer. 2017 Dec 28;17(1):893. doi: 10.1186/s12885-017-3918-9. PMID 29282088
- See also: Related Info — http://www.ikf-nordwest.de/